CLINICAL TRIAL: NCT07406659
Title: Early Effects of Different Inspiratory Muscle Training on Disease Clinical Course, Respiratory Parameters, Functional Capacity and Quality of Life in Patients With COPD
Brief Title: Different Inspiratory Muscle Trainings in Patients With COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, ERDİ KAYABINAR, Assistant Professor, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/432
Record Dates: First submitted 2025-12-17; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Respiratory Muscle Training; Lung Capacities
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Randomised, Controlled, Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Basic Inspiratory Muscle Training (Experimental): The participant will complete IMT training with a physiotherapist one day a week and without a supervisor for the remaining 6 days, 15 minutes in the morning and 15 minutes in the evening.
  Interventions: Other: Basic Inspiratory Muscle Training
- Functional Inspiratory Muscle Training (Experimental): The participant will follow the same Basic IMT program for the first four weeks, and then perform the specified exercises for the remaining four weeks, 3 days a week, for 30 minutes, under the supervision of a physiotherapist. The remaining four days will include 15-minute Basic IMT training in the morning and evening, without a supervisor.
  Interventions: Other: Functional Inspiratory Muscle Training
- Control (Active Comparator): Simple upper extremity exercises and diaphragmatic breathing exercises will be given with equipment suitable for the home environment, 1 day a week accompanied by a physiotherapist for 30 minutes, and the remaining 6 days without a supervisor for 15 minutes in the morning and 15 minutes in the evening. (8-12 repetitions, 2 sets, 1-2 minute break)
  Interventions: Other: Control

INTERVENTIONS:
Other: Basic Inspiratory Muscle Training — The participant will complete IMT training with a physiotherapist one day a week and without a supervisor for the remaining 6 days, 15 minutes in the morning and 15 minutes in the evening.
  Arms: Basic Inspiratory Muscle Training
Other: Functional Inspiratory Muscle Training — Following 4 weeks of Basic IMT, the patient will undergo 30-minute exercises and IMT, three days a week, for 4 weeks, accompanied by a physiotherapist. The patient will continue 15-minute Basic IMT training morning and evening, four days a week, without a supervisor. Exercises will be performed 8-12 times, in 2 sets, with 1-2 minute breaks. Supine chin-up position, lowering and lifting bent legs to the side, Supine chin-up position, 90° hip flexion of one leg, then sliding the heel to extend the knee and 45° straight leg raise, Supine chin-up position, 90° hip flexion of the leg in the chin-up position, Bilateral 90° hip flexion of the legs in the chin-up position, Supine chin-up position, opposite knee extension and shoulder flexion, Cross arm-leg raises in the crawling position, shoulder flexion and extension on mobile surfaces, Back slide on the wall, Lunge by stepping forward, Lifting weight from the floor and lifting it overhead, Bridging, Crunches, Modified push-up
  Arms: Functional Inspiratory Muscle Training
Other: Control — Simple upper extremity exercises and diaphragmatic breathing exercises will be given with equipment suitable for the home environment, 1 day a week accompanied by a physiotherapist for 30 minutes, and the remaining 6 days without a supervisor for 15 minutes in the morning and 15 minutes in the evening. (8-12 repetitions, 2 sets, 1-2 minute break)
  Arms: Control

SUMMARY:
COPD is one of the most life-threatening pulmonary diseases. According to the World Health Organization, it is expected to rise to the third leading cause of death by 2030. Smoking is the most significant contributing factor. COPD reduces lung volumes and causes dyspnea. Over time, respiratory muscle weakness develops, leading to hypercapnia, dyspnea, nocturnal oxygen desaturation, and decreased exercise performance. Pulmonary rehabilitation is the most important component of COPD treatment. Respiratory muscle training should be a mandatory component of the pulmonary rehabilitation program. Combining inspiratory muscle training with functional exercises allows the focus to be on respiratory muscle functions beyond the task of breathing. The purpose of this study was to investigate the effects of Functional Inspiratory Muscle Training on the course of the disease.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a progressive respiratory disease with high mortality and morbidity, although it is preventable and treatable. Environmental and genetic factors, primarily smoking, play a role in the development of the disease. The most common symptom in COPD is dyspnea, which is associated with respiratory muscle dysfunction, hyperinflation, and exercise intolerance. Pulmonary rehabilitation, especially exercise training and respiratory muscle training, is a fundamental component of COPD management.

Inspiratory muscle training (IMT) aims to improve dyspnea, exercise capacity, and quality of life by increasing respiratory muscle strength and endurance. In recent years, Functional Inspiratory Muscle Training (F-IMT) has been developed, focusing on the role of respiratory muscles in postural control and trunk stabilization. However, studies on the effects of F-IMT in individuals with COPD are limited.

The aim of our study was to compare the early-term effects of basic IMT and F-IMT on the disease course in individuals with COPD. In this study, we aim to learn which training is more beneficial for individuals with COPD.

Scope: This is a prospective experimental study. The study will be conducted on total 51 individuals who meet the inclusion criteria. The study population will consist of patients admitted to Yalova Training and Research Hospital.

Inclusion Criteria:

Diagnosed with COPD according to GOLD criteria Not having had an acute exacerbation within the last month Ability to walk independently No communication problems Voluntariness to participate in the study

Exclusion Criteria:

Being in a COPD exacerbation Presence of orthopedic or neurological disease that may interfere with assessment and treatment Presence of uncontrolled hypertension and heart disease Method: The minimum sample size for the study was calculated using the GPower 3.1 program, taking into account the literature, using a 95% confidence interval, 80% power, and an effect size of 0.4823177. Accordingly, the minimum sample size for the study was calculated as 45. Considering the possibility of participant withdrawal, an additional 10% of participants will be recruited. Therefore, the study is planned to include total 51 participants. Participants will be included in the study through invitation and announcement. The study will be conducted with individuals who meet the inclusion criteria. Participants will be divided into three groups: the basic IMT group, the F-IMT group, and the control group, each containing 17 participants.

Data Collection Tools:

Demographic Information, Cognitive Performance: It will be measured using the Standardized Mini Mental Test (SMMT), Dyspnea Assessment (Modified Medical Research Council -mMRC), COPD Assessment Test (CAT), Respiratory Function Test: Measurements are taken with a portable spirometer (Cosmed Pony FX, Cosmed, Rome, Italy) while the patient is in a sitting position, Respiratory Muscle Strength Measurement: Maximal inspiratory and expiratory pressure measurements (MIP-MEP) will be taken, Exercise Capacity Assessment (Six-Minute Walk Test - 6MWT), Peripheral Muscle Strength Measurement: Participants' knee extension and grip strength will be assessed. A hand-held dynamometer (Lafayette Manual Muscle Testing System; Lafayette Instrument Company, Lafayette, Indiana, USA) will be used for knee extension strength, and a Baseline BIMS Digital 5-Position Grip Dynamometer (Baseline Evaluation Instruments, USA) will be used for grip strength, Balance Assessment (Berg Balance Scale-BBS): The BBS is used to assess dynamic balance performance, Core Muscle Assessment: The PRONE test will be performed using the Stabilizer™ (Chattanooga Group Inc., Chattanooga, TN) device, Lower Extremity Endurance Assessment (5-Time Sit-to-Stand Test), Depression Assessment (Beck Depression Inventory - BDI), Assessment of Activities of Daily Living (London Chest Activities of Daily Living Scale - LCADL), Quality of Life Assessment (St. George Respiratory Questionnaire-SGRQ), Fatigue Assessment (COPD and Asthma Fatigue Scale), Physical Activity Level Assessment (International Physical Activity Questionnaire Short Form - UFAA-SF).

Group Training Programs:

Participants will be randomized into three groups: basic IMT, functional IMT (F-IMT), and a control group. This randomization will be conducted through randomizer.org, an open-access randomization website. Participants in both groups will be assessed at the initial meeting and provided with an informed consent form. After completing the initial assessment, they will be informed about the device (in use) and the treatment process. Both groups will receive 8 weeks of treatment. IMT will be applied with a threshold pressure loading device (POWERbreathe Classic Light Resistance, PowerBreath, IMT Technologies Ltd, Birmingham, UK). Patients in both groups will receive training at 40% of the initial measured MIP and a 5-10 second rest break after 10-15 respiratory cycles.

1. Basic IMT group: They will complete IMT training once a week with a physiotherapist for 15 minutes in the morning and 15 minutes in the evening, for the remaining 6 days without a supervisor.
2. F-IMT group: After applying the same Basic IMT program for the first four weeks, the remaining four weeks will be spent 3 days a week with a physiotherapist for 30 minutes, accompanied by the specified exercises. For the remaining four days, they will continue Basic IMT training, unsupervised for 15 minutes in the morning and evening.
3. Control group: Simple upper extremity exercises and diaphragmatic breathing exercises will be performed with equipment suitable for home use, 30 minutes with a physiotherapist once a week, and 15 minutes in the morning and 15 minutes in the evening, unsupervised for the remaining six days. (8-12 repetitions, 2 sets, 1-2 minute break) F-IMT group exercises: Each exercise will be performed simultaneously with the IMT device for 8-12 repetitions, 2 sets. There will be a 1-2 minute break between exercises. -Alternating between lowering and raising bent legs while supine in a chin-up position

   * Alternating between lowering and raising bent legs while supine in a chin-up position
   * Alternating between 90° hip flexion of one leg, then sliding the heel to extend the knee and performing a 45° straight leg raise
   * Alternating between 90° hip flexion of the opposite leg while supine in a chin-up position
   * Alternating between 90° hip flexion of the legs while supine in a chin-up position
   * Contralateral knee extension and shoulder flexion while supine in a chin-up position
   * Crawling cross-leg raises
   * Shoulder flexion and extension on unstable surfaces
   * Back slides on a wall
   * Lunges by stepping forward
   * Lifting a weight from the floor and lifting it overhead while maintaining a neutral spine
   * Bridging exercises
   * Crunches
   * Modified push-ups (Kisner et al., 2017)

ELIGIBILITY:
Inclusion Criteria:

Having a COPD diagnosis according to GOLD criteria Having not had an acute exacerbation within the last month Being able to walk independently Having no communication problems Voluntarily participating in the study

Exclusion Criteria:

Being in a COPD exacerbation Having an orthopedic or neurological disease that would prevent assessment and treatment Having uncontrolled hypertension and heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dyspnea Assessment | Baseline and through study completion, an average of 8 weeks
  Modified Medical Research Council -mMRC: The mMRC used for dyspnea assessment consists of five stages. Stage 0 represents mild dyspnea, and Stage 4 represents severe dyspnea (Bestall et al., 1999).
COPD Assesment Test | Baseline and through study completion, an average of 8 weeks
  COPD Assessment Test (CAT): The test consists of eight questions that examine cough, phlegm, shortness of breath, home and outdoor difficulties, sleep, and fatigue parameters. The maximum score is 40. As the score increases, symptoms worsen. The validity and reliability of the Turkish version was conducted by Yorgancıoğlu et al. (Yorgancioglu, 2012).
Pulmonary Function Testing | Baseline and through study completion, an average of 8 weeks
  Measurements are taken with a portable spirometer (Cosmed Pony FX, Cosmed, Rome, Italy) while the patient is in a seated position. Forced expiratory volume in one second (FEV1) is measured (Miller et al., 2005).
Pulmonary Function Testing | Baseline and through study completion, an average of 8 weeks
  Measurements are taken with a portable spirometer (Cosmed Pony FX, Cosmed, Rome, Italy) while the patient is in a seated position. Forced vital capacity (FVC) is measured (Miller et al., 2005).
Pulmonary Function Testing | Baseline and through study completion, an average of 8 weeks
  Measurements are taken with a portable spirometer (Cosmed Pony FX, Cosmed, Rome, Italy) while the patient is in a seated position. The ratio of forced expiratory volume in one second to forced vital capacity (FEV1/FVC) is measured (Miller et al., 2005).
Pulmonary Function Testing | Baseline and through study completion, an average of 8 weeks
  Measurements are made with a portable spirometer (Cosmed Pony FX, Cosmed, Rome, Italy) with the patient in a sitting position. Peak expiratory flow rate (PEF) are measured (Miller et al., 2005).
Pulmonary Function Testing | Baseline and through study completion, an average of 8 weeks
  Measurements are made with a portable spirometer (Cosmed Pony FX, Cosmed, Rome, Italy) with the patient in a sitting position. Flow rate at 25-75% of forced vital capacity (FEF 25-75%) are measured (Miller et al., 2005).
Pulmonary Function Testing | Baseline and through study completion, an average of 8 weeks
  Measurements are made with a portable spirometer (Cosmed Pony FX, Cosmed, Rome, Italy) with the patient in a sitting position. Vital capacity (VC) are measured (Miller et al., 2005).
Respiratory Muscle Strength Measurement | Baseline and through study completion, an average of 8 weeks
  Maximal inspiratory pressure measurements (MIP) will be taken. For the MIP measurement, the participant sits in a chair and, with a nose clip attached, is asked to take a maximum inspiration through the mouth for 1-3 seconds (Neder et al., 1999)..
Respiratory Muscle Strength Measurement | Baseline and through study completion, an average of 8 weeks
  Maximal expiratory pressure measurements (MEP) will be taken. For the MEP measurement, the participant is asked to take a maximum inspiration and then a maximum expiration for 1-3 seconds. After performing both measurements three times, the best reading is recorded (Neder et al., 1999).
Exercise Capacity Assessment | Baseline and through study completion, an average of 8 weeks
  Six-Minute Walk Test - 6MWT: The six-minute walk test is one of the most frequently used field tests in clinical settings due to its practicality and low cost, assessing submaximal functional capacity. The test is conducted in a 30-meter corridor. After being informed about the test, the participant is asked to walk in a marked area in the corridor for six minutes, and the total distance is recorded. It is recommended that it be performed three times at regular intervals throughout the day, and the best distance recorded. The patient may stop and rest at any time and use assistive devices if available. Blood pressure, heart rate, oxygen saturation, fatigue, and dyspnea are measured before and after the test. In individuals with COPD, a walk of <350 meters is associated with lower exercise capacity and increased mortality risk (Ceylan, 2014). A 6-minute walk will result in a report calculating the total distance walked in meters.

SECONDARY OUTCOMES:
Cognitive Performance | Baseline and through study completion, an average of 8 weeks
  This will be measured with the Standardized Mini Mental Test (SMMT). The Mini Mental Test, developed by Folstein et al., is used to assess an individual's cognitive performance. The maximum score a patient can achieve on the 11-question test, which includes orientation, recording memory, attention and calculation, recall, and language sections, is 30 (Folstein et al., 1975). The higher the score, the better the situation. 0-17 points indicate severe impairment, 18-23 points indicate moderate impairment, 24-26 points indicate mild cognitive impairment, and 27-30 points indicate normal levels (Creavin et al., 2016). The Turkish validity and reliability study was conducted by Güngen et al. (Güngen et al., 2002).
Peripheral Muscle Strength Measurement | Baseline and through study completion, an average of 8 weeks
  Participants' knee extension and grip strength will be assessed. A hand-held dynamometer (Lafayette Manual Muscle Testing System; Lafayette Instrument Company, Lafayette, Indiana, USA) will be used for knee extension strength, and a Baseline BIMS Digital 5-Position Grip Dynamometer (Baseline Evaluation Instruments, USA) will be used for grip strength. Measurements are taken with the participant seated in a chair. Grip strength is measured in the standard position recommended by the American Association of Hand Therapists. Positions include shoulder adduction, forearm neutral position, elbow flexion at 90 degrees, wrist extension at 0-30 degrees, and ulnar deviation of 15 degrees (Tregdet and Davis, 2000). The best value after performing each measurement three times is recorded.
Balance Assessment (Berg Balance Scale-BDI) | Baseline and through study completion, an average of 8 weeks
  The BDI is used to assess dynamic balance performance. It is evaluated under 14 headings, each with a score of 0-4, for a total of 0-56. 56 is the highest score and indicates complete unsupported balance performance. Scores between 0-20 represent high fall risk, 21-40 represent moderate fall risk, and 41-56 represent low fall risk. Its validity and reliability in Turkish were conducted by Şahin et al. (Sahin et al., 2008).
Core Muscle Assessment | Baseline and through study completion, an average of 8 weeks
  The PRONE test will be performed using the Stabilizer™ (Chattanooga Group Inc., Chattanooga, TN) device. Before the test, the patient is instructed to perform an abdominal wall retraction. The device is placed under the abdomen with the patient lying prone. After the manometer pressure is set at 70 mmHg, the patient is asked to perform and maintain the abdominal wall retraction. The test is repeated three times, and the highest value is recorded (de Paula Lima et al., 2011).
Lower Extremity Endurance Assessment (5-Time Sit-to-Stand Test) | Baseline and through study completion, an average of 8 weeks
  The 5-Time Sit-to-Stand Test is an easy-to-administer lower extremity endurance test because it only requires a chair. Patients are asked to sit down and stand up five times in a chair with a backrest and no armrests, without arm support. The total time in seconds is recorded after completing the test (Mong et al., 2010).
Depression Assessment (Beck Depression Inventory-BDI) | Baseline and through study completion, an average of 8 weeks
  The BDI is a scale used to assess depression. It consists of 21 items, each with four options. The scale has a scoring system of 0-3. The lowest score a participant can receive on this scale is 0 and the highest is 63. Higher scores indicate increasing levels of depression. Total scores are divided into 4 groups: 0-9 points: "minimal depression," 10-16 points: "mild depression," 17-29 points: "moderate depression," and 30 points and above: "severe depression." The Turkish reliability study of this scale was conducted by Hisli in 1988 (Hisli, 1989).
Activity of Daily Living Assessment | Baseline and through study completion, an average of 8 weeks
  London Chest Activities of Daily Living Scale - LCADL: There are four subheadings and 15 items, including personal care, housework, physical activity, and leisure time. Each item is scored between 0 and 5. The scale is scored as the total score of the subheadings and the scale. The maximum total score is 75. As the total score increases, so does dependence on activities of daily living (Janaudis-Ferreira et al., 2014). Its validity and reliability in Turkish were conducted by Saka et al.
Quality of Life Assessment | Baseline and through study completion, an average of 8 weeks
  St. George Respiratory Questionnaire-SGRQ: This questionnaire is used to measure health-related quality of life in individuals with respiratory diseases. It consists of 50 items in three sections: symptoms, activities, and disease effects. Scoring ranges from 0 to 100, with higher scores indicating worsening health status. The validity and reliability of the scale was conducted by Polatlı et al. (Polatlı et al., 2013).
Fatigue Assessment | Baseline and through study completion, an average of 8 weeks
  COPD and Asthma Fatigue Scale: This is a 12-item scale specifically developed for the assessment of fatigue in patients with COPD and asthma. Questions are on a five-point Likert-type scale, yielding a score between 12 and 60. The scale score is calculated out of 100 using the formula: Scale score = [(Total Raw Score-12 /48) x 100]. A higher score indicates greater fatigue (Revicki et al., 2010). The Turkish validity and reliability were made by Aslan and Öztunç (Aslan and Öztunç, 2013).
Physical Activity Level Assessment | Baseline and through study completion, an average of 8 weeks
  Short Form of the International Physical Activity Questionnaire-IPAQ-SF: This questionnaire, whose validity and reliability in Turkish were developed by Sağlam et al., consists of 7 questions. It asks about vigorous and moderate physical activities, including walking and sitting activities, performed within the last week, on how many days per week and for how long. Sitting activity is not included in the scoring section (Sağlam et al., 2010). MET values of the activities were used as 8 METs for vigorous physical activities, 4 METs for moderate physical activities, and 3.3 METs for walking, and the total score was recorded as MET-min/week. The total duration (minutes) and frequency (days) of each are required for score calculation. The MET score is obtained by multiplying the MET value of the activity by the number of days and minutes. The results are evaluated in three categories: inactive, moderately active, and active: Inactive, Moderately active, Active (Craig et al., 2003).

CONTACTS AND LOCATIONS:
Overall Officials: Erdi KAYABINAR, PhD, Principal Investigator — University of Yalova
Locations (1):
- Yalova University, Yalova, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ammous O, Feki W, Lotfi T, Khamis AM, Gosselink R, Rebai A, Kammoun S. Inspiratory muscle training, with or without concomitant pulmonary rehabilitation, for chronic obstructive pulmonary disease (COPD). Cochrane Database Syst Rev. 2023 Jan 6;1(1):CD013778. doi: 10.1002/14651858.CD013778.pub2. PMID 36606682
- [Background] Beaumont M, Mialon P, Le Ber C, Le Mevel P, Peran L, Meurisse O, Morelot-Panzini C, Dion A, Couturaud F. Effects of inspiratory muscle training on dyspnoea in severe COPD patients during pulmonary rehabilitation: controlled randomised trial. Eur Respir J. 2018 Jan 25;51(1):1701107. doi: 10.1183/13993003.01107-2017. Print 2018 Jan. PMID 29371379
- [Background] Ekren, P. K., Gürgün, A. 2013. "KOAH'da pulmoner rehabilitasyon: kime, ne zaman, nasıl", Güncel Göğüs Hastalıkları Serisi, 1(1), 124-35.
- [Background] Ergün, P. 2019. "Pulmoner rehabilitasyon güncel yaklaşımlar" Güncel Göğüs Hastalıkları Serisi, 7, 7-18.
- [Background] Firat, M., Saglam, M., Calik-Kutukcu, E., Inal-Ince, D., Ardali-Duzgun, S., Yildirim, T., Vardar-Yagli, N. 2024. Effect of functional inspiratory muscle training in chronic kidney disease", Eur Respir J, 64, 68.
- [Background] Gezgen, A., Erk, M., Müsellim, B., Demir, T., Mutlu, B. 2001. "KOAH'da Üst Ekstremite Egzersizlerinin Yaşam Kalitesine ve Solunum Fonksiyonlarına Etkisi", Solunum Dergisi, 3, 60-65.
- [Background] Global Initiative For Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease. Revised 2011.
- [Background] Gökçek, Ö., Doğru Hüzmeli, E., Katayıfçı, N. 2019. "Kronik obstrüktif akciğer hastalarında dispnenin yaşam kalitesi ve depresyona etkisi", ACU Sağlık Bil Dergisi, 10(1), 84-88.
- [Background] Han B, Chen Z, Ruan B, Chen Y, Lv Y, Li C, Yu L. Effects of Inspiratory Muscle Training in People with Chronic Obstructive Pulmonary Disease: A Systematic Review and Meta-Analysis. Life (Basel). 2024 Nov 12;14(11):1470. doi: 10.3390/life14111470. PMID 39598268
- [Background] Huzmeli I, Katayifci N, Abay B, Akkus O, Ozer AY. The effectiveness of functional inspiratory muscle training on exercise capacity and peripheral muscle strength in patients with essential hypertension: a three-arm randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Feb 28;17(1):29. doi: 10.1186/s13102-025-01082-w. PMID 40022256
- [Background] İnce, D., Savcı, S., Sağlam, M., Arıkan, H., Çöplü, L. 2011. "Kronik obstrüktif akciğer hastalarında sigara öyküsü ve fonksiyonel kapasite arasındaki ilişki", Fizyoterapi Rehabilitasyon, 22(1), 39-43
- [Background] Keskin, T., Başkurt, Z. 2021. "KOAH Tanılı Yaşlı Bireylerde Pulmoner Rehabilitasyon", Celal Bayar Üniversitesi Sağlık Bilimleri Enstitüsü Dergisi, 8(1), 157-161.
- [Background] Li Z, Liu S, Wang L, Smith L. Mind-Body Exercise for Anxiety and Depression in COPD Patients: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2019 Dec 18;17(1):22. doi: 10.3390/ijerph17010022. PMID 31861418
- [Background] McConnell, A. 2013. Respiratory Muscle Training, Theory and Practice, Edinburg: Elsevier.
- [Background] Özdemir, F., Koca, T., Berber, N., Şahin, Ş. 2018. "Astım ve KOAH Hastalarının Fiziksel Aktivite Düzeylerinin Değerlendirilmesi", KSÜ Tıp Fakültesi Dergisi, 14(1), 20-23.
- [Background] Ozsoy I, Kahraman BO, Ozsoy G, Ilcin N, Tekin N, Savci S. Effects of an Integrated Exercise Program Including "Functional" Inspiratory Muscle Training in Geriatric Individuals with and without Chronic Obstructive Pulmonary Disease. Ann Geriatr Med Res. 2021 Mar;25(1):45-54. doi: 10.4235/agmr.21.0014. Epub 2021 Mar 30. PMID 33794587
- [Background] Özyılmaz, S., Gürses, H. N. 2012. "KOAH'ta Göğüs Fizyoterapisi". KOAH'ta pulmoner rehabilitasyon. Editörler: Gürses HN, Biber Ç. TÜSAD Eğitim Kitapları Serisi. İstanbul: Probiz Ltd Şti.
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Pesci A, Balbi B, Majori M, Cacciani G, Bertacco S, Alciato P, Donner CF. Inflammatory cells and mediators in bronchial lavage of patients with chronic obstructive pulmonary disease. Eur Respir J. 1998 Aug;12(2):380-6. doi: 10.1183/09031936.98.12020380. PMID 9727789
- [Background] Saetta M, Di Stefano A, Maestrelli P, Ferraresso A, Drigo R, Potena A, Ciaccia A, Fabbri LM. Activated T-lymphocytes and macrophages in bronchial mucosa of subjects with chronic bronchitis. Am Rev Respir Dis. 1993 Feb;147(2):301-6. doi: 10.1164/ajrccm/147.2.301. PMID 8430952
- [Background] Şahin, H., Pehlivan, E. 2022. "KOAH'da Pulmoner Rehabilitasyon". Kronik Obstrüktif Akciğer Hastalığı (KOAH). Ankara: Dünya Tıp Kitapevi.
- [Background] Saka S, Gurses HN, Bayram M. Effect of inspiratory muscle training on dyspnea-related kinesiophobia in chronic obstructive pulmonary disease: A randomized controlled trial. Complement Ther Clin Pract. 2021 Aug;44:101418. doi: 10.1016/j.ctcp.2021.101418. Epub 2021 May 14. PMID 34034036
- [Background] Troosters T, Janssens W, Demeyer H, Rabinovich RA. Pulmonary rehabilitation and physical interventions. Eur Respir Rev. 2023 Jun 7;32(168):220222. doi: 10.1183/16000617.0222-2022. Print 2023 Jun 30. PMID 37286219
- [Background] Tütüneken, YE. (2024), "Kronik İnmeli Hastalarda İnspiratuar Kas Eğitimine Karşı Fonksiyonel İnspiratuar Kas Eğitiminin Gövde Kontrolüne ve Solunum Fonksiyonlarına Etkisi''
- [Background] Yüksel, E. G., Ursavaş, A., Irdesel, J., Koç, M., Uzaslan, E. K., Güneş, S., Özyardimci, N. 2005. "Kronik Obstrüktif Akciğer Hastaliğinda Multidisipliner Pulmoner Rehabilitasyon Programinin Etkinliği", Turkiye Klinikleri Archives of Lung, 6(3), 115-119.
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] Yorgancioglu A, Polatli M, Aydemir O, Yilmaz Demirci N, Kirkil G, Nayci Atis S, Kokturk N, Uysal A, Akdemir SE, Ozgur ES, Gunakan G. [Reliability and validity of Turkish version of COPD assessment test]. Tuberk Toraks. 2012;60(4):314-20. doi: 10.5578/tt.4321. Turkish. PMID 23289460
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550
- [Background] Ceylan, E. (2014). Kardiyopulmoner egzersiz testleri. Journal of Clinical and Experimental Investigations, 5(3), 504-509.
- [Background] Tredgett MW, Davis TR. Rapid repeat testing of grip strength for detection of faked hand weakness. J Hand Surg Br. 2000 Aug;25(4):372-5. doi: 10.1054/jhsb.2000.0433. PMID 11058007
- [Background] Sahin F, Yilmaz F, Ozmaden A, Kotevolu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Berg Balance Scale. J Geriatr Phys Ther. 2008;31(1):32-7. doi: 10.1519/00139143-200831010-00006. PMID 18489806
- [Background] de Paula Lima PO, de Oliveira RR, Costa LO, Laurentino GE. Measurement properties of the pressure biofeedback unit in the evaluation of transversus abdominis muscle activity: a systematic review. Physiotherapy. 2011 Jun;97(2):100-6. doi: 10.1016/j.physio.2010.08.004. Epub 2010 Oct 23. PMID 21497243
- [Background] Mong Y, Teo TW, Ng SS. 5-repetition sit-to-stand test in subjects with chronic stroke: reliability and validity. Arch Phys Med Rehabil. 2010 Mar;91(3):407-13. doi: 10.1016/j.apmr.2009.10.030. PMID 20298832
- [Background] HİSLİ, N. (1989). "Beck Depresyon Envanterinin üniversite öğrencileri için geçerliği, güvenirliği", Psikoloji dergisi, cilt 7, sayi 23, ss. 3-13.
- [Background] Saka S, Savci S, Kutukcu EC, Saglam M, Yagli NV, Ince DI, Guclu MB, Ozalp O, Arikan H, Karakaya G, Coplu L. Validity and Reliability of the Turkish Version of the London Chest Activity of Daily Living Scale in Obstructive Lung Diseases. Turk Thorac J. 2020 Mar 1;21(2):116-121. doi: 10.5152/TurkThoracJ.2019.18155. Print 2020 Mar. PMID 32203002
- [Background] Janaudis-Ferreira T, Beauchamp MK, Robles PG, Goldstein RS, Brooks D. Measurement of activities of daily living in patients with COPD: a systematic review. Chest. 2014 Feb;145(2):253-271. doi: 10.1378/chest.13-0016. PMID 23681416
- [Background] Polatli M, Yorgancioglu A, Aydemir O, Yilmaz Demirci N, Kirkil G, Atis Nayci S, Kokturk N, Uysal A, Akdemir SE, Ozgur ES, Gunakan G. [Validity and reliability of Turkish version of St. George's respiratory questionnaire]. Tuberk Toraks. 2013;61(2):81-7. doi: 10.5578/tt.5404. Turkish. PMID 23875584
- [Background] Revicki DA, Meads DM, McKenna SP, Gale R, Glendenning GA, Pokrzywinski MHA. COPD and asthma fatigue scale (CAFS): development and psychometric assessment. Health Outcomes Res Med 2010; 1(1): 5-16.
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Kisner, C., Colby, L. A., & Borstad, J. (2017). Therapeutic exercise: foundations and techniques. Fa Davis.
- [Background] Creavin ST, Wisniewski S, Noel-Storr AH, Trevelyan CM, Hampton T, Rayment D, Thom VM, Nash KJ, Elhamoui H, Milligan R, Patel AS, Tsivos DV, Wing T, Phillips E, Kellman SM, Shackleton HL, Singleton GF, Neale BE, Watton ME, Cullum S. Mini-Mental State Examination (MMSE) for the detection of dementia in clinically unevaluated people aged 65 and over in community and primary care populations. Cochrane Database Syst Rev. 2016 Jan 13;2016(1):CD011145. doi: 10.1002/14651858.CD011145.pub2. PMID 26760674
- [Background] Arslan, S. ve Öztunç, G. (2013). Kronik Obstrüktif Akciğer Hastalığı ve Astım Yorgunluk Ölçeği'nin geçerlilik ve güvenirliği. Hemşirelikte Araştırma Geliştirme Dergisi, 15(1), 48-60.